CLINICAL TRIAL: NCT05606042
Title: Curvafix® Intramedullary System for Fixation of Pelvic and Acetabular Fractures, A Post Market Performance Evaluation
Brief Title: Curvafix® Intramedullary System for Fixation of Pelvic and Acetabular Fractures, A Post Market Evaluation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CurvaFix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-0002; ACTRN12622001125718 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Pelvic Ring Fracture; Acetabular Fracture; Pelvic Fracture; Pelvic Fracture Acetabulum
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- IM Implant: Male and female patients who present with a pelvic ring and/or acetabular fracture that has recently undergone surgery to be fixed with a CurvaFix IM Implant.
  Interventions: Device: IM Implant

INTERVENTIONS:
Device: IM Implant — Patients that have had surgical interventions with one or more IM Implant as part of standard of care for a pelvic and/or acetabular fracture

SUMMARY:
Prospective, single arm, post-market evaluation to evaluate the use and performance of the IM Implant in a post market setting.

DETAILED DESCRIPTION:
This study will evaluate the use and performance of the Curvafix IM intramedullary system for pelvic fixation in a post-market setting. Study participants will undergo follow-up care per institutional practice and data will then be collected from participant medical records. There will be no active patient participation requirements outside of standard of care. Any follow up evaluations will be documented and reported through 6 months post-implantation. The study will evaluate secondary surgical interventions as a primary study endpoint. Data will also be collected and analyzed for pelvic reduction stability, fracture healing, participant mobility/ambulation, and general health economics.

ELIGIBILITY:
Inclusion Criteria:

* Subject, or their Authorized Representative, is willing and able to provide written informed consent, including authorization to release health information
* Subject has undergone pelvic or acetabular fixation using the IM Implant and the IM Implant was placed according to the manufacturer's labeling.
* Subject's pelvic or acetabular fixation with the IM Implant occurred within the last 30 calendar days.

Exclusion Criteria:

* Subject is unwilling or unable to provide written informed consent and/or does not have an authorized representative who can provide consent on their behalf
* Subject presents with any condition or situation which, in the Investigator's opinion, puts the Subject at risk, could confound the study results, or may interfere with the Subject's participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected from medical facility study sites that have agreed to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Secondary Surgical Interventions (SSIs) | 6 months post-implantation
  Performance will be evaluated based upon the number of Secondary Surgical Interventions (SSIs) that occur within the subject's participation as identified through a review of subject medical records.

SECONDARY OUTCOMES:
Mobility | 6 months post-implantation
  Mobility (ability to advance to weight bearing) assessed by medical record review
Pelvic Reduction Stability | 6 months post-implantation
  Pelvic reduction stability (ability to maintain reduction over time) assessed by medical record review
Health Economics | 6 months post-implantation
  General health economics (length of hospital stay) assessed by medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hebert, Study Director — Clin-Assist, LLC
Locations (4):
- United States (4):
  - Memorial Medical Center, Springfield, Springfield, Illinois
  - Missouri Orthopaedic Institute, Columbia, Missouri
  - Mount Carmel Research Institute, Columbus, Ohio
  - UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No